CLINICAL TRIAL: NCT06292325
Title: Psychological Aspects in Modifying Apnea/Hypopnea Indices and Nadir of Saturation in Obstructive Sleep Apnea Syndrome (OSA)
Brief Title: Psychological Aspects in OSA
Acronym: PSICOSA
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Eleonora Volpato, Clinical Professor, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: FDG_88-17
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Osa Syndrome
Keywords: Quality of life; Couple Relationship Quality; CPAP; Sleep Apnea; Sleep Disturbance; Adherence to treatment
MeSH Terms: conditions — Carnevale syndrome; Sleep Apnea Syndromes; Parasomnias; Treatment Adherence and Compliance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) — CPAP is the gold standard therapy for Obstructive Sleep Apnea. It consists of a machine that delivers a constant and steady air pressure through a mask worn over the nose or both nose and mouth during sleep. This continuous flow of air helps to keep the airway open, preventing episodes of airway collapse and obstruction characteristic of OSA. CPAP therapy is highly effective in reducing symptoms such as snoring, daytime sleepiness, and fatigue, as well as improving overall sleep quality and decreasing the risk of complications associated with untreated OSA, such as cardiovascular issues. It is considered the gold standard treatment for moderate to severe OSA and is often prescribed after a sleep study confirms the diagnosis. CPAP machines come in various designs and features to suit individual needs and preferences, and proper adjustment and compliance are essential for optimal treatment outcomes.

SUMMARY:
The research project consists of an observational study. Obstructive Sleep Apnea (OSA) is a condition characterized by recurrent episodes of upper airway collapse during sleep, leading to decreased blood oxygen levels and disruptions of normal sleep patterns. Estimates of its prevalence vary, but its impact on patients' quality of life is evident.

Through a qualitative analysis (semi-structured interviews for both patients and bed partners) and a quantitative analysis (APIM Model), this research aims to explore the perception and awareness of the disease and its impact on the individual and couple's lives of patients with OSA and their bed partners, to assess patients' perceptions of the disease, illness management (CPAP experience) and symptoms, as well as their bed partners' perceptions. Moreover, psychological aspects of living with OSA, such as perceived stress, depression, anxiety, sleep quality, daily sleepiness will be studied to observe the association with Continuous Positive Airway Pressure (CPAP) adherence.

DETAILED DESCRIPTION:
Firstly, a series of semi-structured interviews will be conducted with patients with OSA, at different levels of CPAP adaptation as well as with bed partners of patients who are experiencieng CPAP treatment with OSA.

After that, a quantitative analysis will be conducted to explore dyadic dynamics between patients with OSA and their bed partners.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatient patients
* over 18 years of age
* Diagnosis of Obstructive Sleep Apnea Syndrome
* Absence of cognitive impairments
* Having a bedpartner

Exclusion Criteria:

* Oncological comorbidities
* Dementia, as reported in the medical record
* Ongoing treatment with phosphodiesterase-5 inhibitors, hypogonadism, or severe lung diseases
* Exacerbations requiring hospitalization or the use of corticosteroids and antibiotics in the last two months
* Lack of consent
* Lack of a bedpartner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult OSA patients already adapted to CPAP therapy or who have just started adaptation to CPAP, with any severity level of disease and their bedpartners. So the study will include both the partners (Dyads).
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Brief Illness Perception Questionnaire (Brief IPQ) | from May 2023 to May 2024
  It is a self-administered questionnaire consisting of nine items rated on a scale of 0-10. The first five items assess cognitive perceptions such as the impact on life (item 1); duration of illness (item 2); disease control (item 3); beliefs about treatment effectiveness (item 4); and symptom experience (item 5). Items 6 and 8 assess emotional aspects, such as concern about the illness and mood. Item 7 assesses the level of understanding of the illness. The last item requires respondents to rank the three factors that caused the illness. Cut-offs for the total score are determined as follows: <42 indicates a mild threat, 42-49 indicates a moderate threat, and ≥50 indicates a high threat.
CPAP therapy adherence (hours/night) | from May 2023 to May 2024
  CPAP therapy average daily adherence will be evaluated through data extraction from the integrated ventilator software during hospital visits.
Dyadic Adjustment Scale (DAS) | from May 2023 to May 2024
  A self-administered questionnaire consisting of 32 items divided into 4 subscales: "Consensus on important issues," "Satisfaction with relationship status," "Doing things together," and "Satisfaction with emotional and sexual life." To obtain the interpretation of the questionnaire, the average score for each area is calculated, noting that in the responses to questions 30 and 31, the corresponding score is 0 for NO and 1 for YES.

SECONDARY OUTCOMES:
The experience in close relationships-revised (ECR-R) Scale | from May 2023 to May 2024
  It is a self-administered questionnaire, consisting of two subscales of 18 items each, which assess Avoidance and Anxiety related to attachment in relationships with romantic partners. The items are rated on a 7-point Likert scale (1=strongly disagree; 7=strongly agree), with higher scores indicating greater attachment avoidance and anxious attachment with romantic partners.
The Psychological General Well-Being Index (PGWB-S) | from May 2023 to May 2024
  The short version with 6 items of the self-administered questionnaire composed of 22 items, which provides a subjective assessment of one's psychological well-being, on a 6-step Likert scale (0-5). Higher scores indicate greater psychological well-being.
The Patient Health Questionnaire - 9 (PHQ-9) | from May 2023 to May 2024
  It consists of 9 items corresponding to symptoms of major depression according to the DSM-IV. Scores range from 0 to 27. Scores between 0 and 9 indicate subthreshold depression. A score of 10 is identified as the point where the sensitivity and specificity of the instrument are recognized as optimal for detecting clinically significant depression.
The Generalized Anxiety Scale -7 (GAD-7) | from May 2023 to May 2024
  It's a 7 items scale, designed to assess the severity of generalized anxiety disorder symptoms. Comprising seven items that inquire about common anxiety symptoms such as feeling nervous, worrying excessively, and experiencing restlessness. Each item on the scale is scored on a Likert scale ranging from 0 to 3, with responses indicating the frequency of symptoms over the past two weeks. The total score ranges from 0 to 21, with higher scores indicating greater severity of anxiety symptoms.
The Mannheim Dream Questionnaire (MADRE) | from May 2023 to May 2024
  It is a 21-items scale used to explore dream content on a 7-point Likert scale, from 0 (never) to 6 (almost every morning). It consists of a series of structured questions aimed at investigating various aspects of the dream experience.
The EP worth scale (ESS) | from May 2023 to May 2024
  A self-administered questionnaire, consisting of 8 items, on a 4-step Likert scale (0-3), regarding usual lifestyle habits in the recent period, aimed at exploring the presence of daytime sleepiness. Scores ≥10 indicate excessive daytime sleepiness.
Pittsburgh Sleep Quality Index (PSQI) | from May 2023 to May 2024
  A self-administered tool consisting of 19 items that assesses sleep quality. Patients can be classified as High Risk (if there are 2 or more categories in which the score is positive) or Low Risk (if there are no categories present or only one in which the score is positive), based on their responses to individual items and their overall scores in symptom categories; in addition, the 5 questions intended for the bed partner will also be included.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parish JM, Lyng PJ. Quality of life in bed partners of patients with obstructive sleep apnea or hypopnea after treatment with continuous positive airway pressure. Chest. 2003 Sep;124(3):942-7. doi: 10.1378/chest.124.3.942. PMID 12970021
- [Background] Batool-Anwar S, Goodwin JL, Kushida CA, Walsh JA, Simon RD, Nichols DA, Quan SF. Impact of continuous positive airway pressure (CPAP) on quality of life in patients with obstructive sleep apnea (OSA). J Sleep Res. 2016 Dec;25(6):731-738. doi: 10.1111/jsr.12430. Epub 2016 May 30. PMID 27242272
- [Background] Sawyer AM, Gooneratne NS, Marcus CL, Ofer D, Richards KC, Weaver TE. A systematic review of CPAP adherence across age groups: clinical and empiric insights for developing CPAP adherence interventions. Sleep Med Rev. 2011 Dec;15(6):343-56. doi: 10.1016/j.smrv.2011.01.003. Epub 2011 Jun 8. PMID 21652236
- [Background] Chu, C. M., Wu, S. Y., Yu, C. C., & Huang, C. Y. (2021). Sleep Disturbance and Depressive Tendency in Bed Partners of Patients With Obstructive Sleep Apnea.